CLINICAL TRIAL: NCT05533307
Title: Mediolateral Episiotomy in Nulliparous Women Increases the Risk of Sexual Dysfunction
Status: Completed | Type: Observational
Sponsor: Batman Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erhan Okuyan,M.D, M.D,Obstetric and gynecology division, Batman Training and Research Hospital
Other Study IDs: EOkuyan
Record Dates: First submitted 2022-09-03; First posted 2022-09-09 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Episiotomy; Complications
Keywords: sexuel dysfunction; mediolateraş episiotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- nulliparous women with normal birth (not needed mediolateral episitomy)/1: group without mediolateral episiotomy
  Interventions: Diagnostic Test: observational analysis of mediolateral episiotomy with arizona sexuel function scoring after 3 months of normal vaginal birth
- nulliparous women with normal birth (with mediaolateral episiotomy)/2: group with mediolateral episiotomy
  Interventions: Diagnostic Test: observational analysis of mediolateral episiotomy with arizona sexuel function scoring after 3 months of normal vaginal birth

INTERVENTIONS:
Diagnostic Test: observational analysis of mediolateral episiotomy with arizona sexuel function scoring after 3 months of normal vaginal birth — ASEX (ARİZONA SEXUEL FONCTİON SCORİNG) TEST

SUMMARY:
Postpartum sexual functions may be affected in women who have had a vaginal delivery by performing an episiotomy. The aim of this study is to compare the frequency of sexual dysfunction between women who were delivered with a mediolateral episiotomy and those who were delivered without an episiotomy.

Materials and Methods: A total of 179 women who gave birth in a tertiary center were included in the prospective study. The patients were divided into two groups as women with and without mediolateral episiotomy. The groups were compared in terms of age, body mass index, educational status, and hospitalization time for delivery and Arizona sexual experiences scale (ASEX).

DETAILED DESCRIPTION:
All patients were called up for a control in 6th month after delivery and sexual funciton was evaluated according to The Arizona Sexual Experience Scale (ASEX). In our study, we used the ASEX test, age, education level, BMI and time spent in hospital for delivery to investigate sexual dysfunction in healthy women who had a vaginal delivery with or without mediolateral episiotomy. The ASEX test is a 5-question survey. In the questionnaire, women were questioned for sexual drive, arousal, vaginal lubrication, ability to reach orgasm, satisfaction from the orgasm. Women gave points from 1 to 6 and their results were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women who gave birth at term
* No smoking or alcohol consumption
* Chronic illness
* Spontaneous labor( The labor was defined as cervical dilatation of at least 2cm with at least 80% of effacement with regular contractions or 4cm dilatation with any effacement with regular contractions or the flow of amniotic fluid.

Exclusion Criteria:

* Exclusion criteria were need of labor induction,
* history of any pregnancy complication (gestational diabetes, hypertension, oligohydramnios, any suspicion of infection or chorioamnionitis…etc.),
* history of multiparity,
* history of sexual dysfunction,
* history of vaginal surgery and frequent vaginal infection.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — nulliparous women with normal vginal birth
Study Population: Nulliparous women who gave birth with or without mediolateral episiotomy at Batman training and research hospital will noted individually. After 3 months of birth all included patients will have an ASEX test for sexuel dysfunction analyse.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of sexuel dysfunction with ASEX(Arizona sexuel fonction scoring) | Sexuel dysfuntion scores after 6 months of normal vaginal birth
  In this study, we prospectively evaluated patients in active labor using ASEX and wanted to investigate the effect of mediolateral episiotomy on female sexual life. Maximum score of Asex scoring is 24 and minimum score is 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Batman Training and Research Hospital, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No